CLINICAL TRIAL: NCT05411367
Title: A Multicenter, Randomized, Double-masked and Placebo-controlled Study Evaluating the Efficacy and Safety of SI-614 Ophthalmic Solution in Patients With Dry Eye
Brief Title: A Study for Evaluation of the Efficacy and Safety of SI-614 Ophthalmic Solution in Patient With Dry Eye
Acronym: SIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Collaborators: ORA, Inc. (Industry); Statistics & Data Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 614/1132
Record Dates: First submitted 2022-06-05; First posted 2022-06-09 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SI-614 (Experimental): One drop of study drug was instilled in each eye 4 times daily for 84 days
  Interventions: Drug: SI-614
- Placebo (Placebo Comparator): One drop of study drug was instilled in each eye 4 times daily for 84 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SI-614 — One drop of study drug was instilled in each eye 4 times daily for 84 days
  Other Names: Chemically modified sodium hyaluronate
  Arms: SI-614
Drug: Placebo — One drop of study drug was instilled in each eye 4 times daily for 84 days
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SI-614 ophthalmic solution compared with placebo in patients with dry eye

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-masked study designed to evaluate the efficacy and safety of SI-614 ophthalmic solution compared to placebo in patients with dry eye. Approximately 230 male and female patients at least 18 years of age with dry eye in both eyes will be randomized to receive treatment with SI-614 or placebo in a 1:1 ratio.

Randomized subjects received assigned study drug bilaterally four times daily. For efficacy endpoints, one "study eye" were defined for each patient based on the criteria at baseline and used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Have history of dry eye in both eyes for at least 6 months prior to Visit 1.
* Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to Visit 1.
* If a female of childbearing potential, have a negative urine pregnancy test at Visit 1 and will be using an adequate method of birth control throughout the study period.

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 or Visit 2, including active blepharitis, meibomian gland dysfunction, lid margin inflammation or ocular allergies that requires therapeutic treatment and/or, in the opinion of the investigator, may interfere with the study parameters.
* Be diagnosed with an ongoing ocular infection (bacterial, viral or fungal), or active ocular inflammation (eg, follicular conjunctivitis) at Visit 1 or Visit 2.
* Have had any ocular surgical procedure within 12 months prior to Visit 1, or have any scheduled ocular surgical procedure during the study period.
* Be a female who is pregnant, nursing an infant, or planning a pregnancy.
* Have a known allergy and/or sensitivity to the study drug or its components.
* Have a condition or is in a situation that, in the opinion of the investigator, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patients' participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Ousler, Study Director — ORA, Inc.
Locations (6):
- United States (6):
  - Eye Research Foundation, Newport Beach, California
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Andover Eye Associates, Inc., Andover, Massachusetts
  - Center for Sight, Henderson, Nevada
  - CORE Inc, Vita Eye Clinic, Shelby, North Carolina
  - Total Eye Care, PA, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a study in which whole participants, not eyes were assigned to Arms/Groups. Patients were randomized to receive treatment with SI-614 or placebo in a 1:1 ratio, and the randomized subjects received assigned study drug bilaterally four times daily. For efficacy endpoints, one "study eye" was defined for each patient at baseline and used for analysis. Therefore, whole patients are assigned to Arms/Groups
Pre-assignment Details: Of the screened 470 subjects, 238 subjects were screen failed, and 232 subjects were randomized (114 subjects in SI-614 and 118 subjects in Placebo).
  From the 232 subjects, 231 subjects (114 subjects in SI-614, and 117 subjects in Placebo) received at least one dose of study drug and 1 subject did not receive study drug.
  Efficacy was analyzed on all randomized subjects (232 subjects). Safety was analyzed on all subjects who receive at least 1 dose of randomized study drug (231 subjects).
Period: Overall Study
Arm/Group | SI-614 | Placebo
Started | 114 | 118
Completed | 100 | 107
Not Completed | 14 | 11
Not completed — Adverse Event | 9 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Administrative Reasons | 2 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Inclusion Criteria Not Met | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SI-614 | Placebo | Total
Number analyzed (Participants) | 114 | 118 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.81) | 64.4 (12.08) | 64.0 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 84 | 166
  Male | 32 | 34 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Race : American Indian or Alaska Native | 0 | 2 | 2
  Race : Asian | 4 | 5 | 9
  Race : Black or African American | 17 | 26 | 43
  Race : Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race : White | 92 | 85 | 177
  Race : Other | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Ethnicity : Hispanic or Latino | 10 | 7 | 17
  Ethnicity : Not Hispanic or Latino | 104 | 111 | 215
Corneal Fluorescein Staining Score [Mean (Standard Deviation); unit: units on a scale] — The examiner instilled sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. After 3-5 minutes after instillation, the staining was graded with a scale, which was a 0 to 4 scale and where grade 0 = No Staining and 4 = Confluent Staining. Higher numbers indicate worse outcome.
  The total score was derived using the sum of the 3 regions such that possible scores range from 0 to 12. Corneal Fluorescein Staining Score were summarized for the study eye.
  units on a scale | 4.54 (1.260) | 4.22 (1.124) | 4.38 (1.201)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 29 in Corneal Fluorescein Staining Score in the Study Eye
Description: The examiner instilled sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. After 3-5 minutes after instillation, the staining was graded with a scale, which was a 0 to 4 scale and where grade 0 = No Staining and 4 = Confluent Staining. Higher numbers indicate worse outcome.
  The total score was derived using the sum of the 3 regions such that possible scores range from 0 to 12.
  For efficacy endpoints, one "study eye" were defined for each patient based on the criteria at baseline and used for analysis. Analyses were for the study eye only.
  Efficacy was analyzed on all randomized subjects (232 subjects: 114 subjects in SI-614 and 118 subjects in Placebo).
Time Frame: 29 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SI-614 | Placebo
Number analyzed (Participants) | 114 | 118
score on a scale | 2.19 (0.182) | 2.31 (0.177)
Statistical Analysis 1: Comparison: SI-614 vs Placebo; Test type: Superiority; p = 0.315, ANCOVA; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.62 to 0.38]

2. Secondary Outcome: Change From Baseline in the Average Score of Ocular Discomfort and Dryness at the Bedtime Assessment From the Patient Daily Diary During Day 1 Through Day 14
Description: Subjects graded the severity of their dry eye disease symptoms in their diary with rating the severity of 5 symptoms. Each symptom rating ranged from 0 to 5 using whole numbers, where 0 = None and 5 = Worst. Higher numbers indicate worse symptomology.
  The average score of the two symptoms of ocular discomfort (where 0 = None and 5 = Worst) and dryness (where 0 = None and 5 = Worst) was measured.
Time Frame: 14 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SI-614 | Placebo
Number analyzed (Participants) | 114 | 118
score on a scale | -0.04 (0.039) | -0.04 (0.039)
Statistical Analysis 1: Comparison: SI-614 vs Placebo; Test type: Superiority; p = 0.487, Mixed Models Analysis; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.11 to 0.11], Standard Error of Mean 0.055

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | SI-614 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/117
Serious Adverse Events (participants affected / at risk) | 4/114 | 3/117
Other Adverse Events (participants affected / at risk) | 31/114 | 23/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SI-614 (N=114) | Placebo (N=117)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SI-614 (N=114) | Placebo (N=117)
Instillation site pain (General disorders) | 21 | 18
Visual acuity reduced (Eye disorders) | 4 | 1
COVID-19 (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator must receive prior, written consent from Sponsor before publishing or presenting the results of the Study

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT05411367/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT05411367/SAP_001.pdf